CLINICAL TRIAL: NCT04285424
Title: Fecal Microbiota Transplantation for Treatment of Steroid Resistant Acute Graft Versus Host Disease of the Gut
Brief Title: FMT for Steroid Resistant Gut Acute GVHD
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Collaborators: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMT-GVHD-7182122
Record Dates: First submitted 2020-02-20; First posted 2020-02-26 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Stem Cell Transplant Complications; Acute Graft-Versus-Host Disease; Fecal Microbiota Transplantation
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HSCT patients with acute steroid-resistant GI-related GVHD (Experimental): Patients will receive 500ml fecal microbiota which were sprayed evenly on the entire colon through colonscopy or duodenal nutrition tube injection which collected from one unrelated healthy donors. Patients receiving FMT treatment will be followed for at least 1,3,5,7 days.Stool, blood and colonic mucosa samples will be serially collected and tested (before pre-treatment, 1,3,5,7 days after FMT).
  Interventions: Biological: Fecal Microbiota Transplantation

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation — The fecal collection produced from a single healthy donor, unrelated to the patients

SUMMARY:
The study aims to evaluate the safety and efficacy of fecal microbiota transplantation (FMT) for the treatment of steroid resistant graft-versus-host-disease (GVHD) of the gut. This strategy might offer a safe and effective therapeutic approach for these patients with a poor prognosis and limited therapeutic options.

DETAILED DESCRIPTION:
Graft-versus-host-disease (GVHD) is a major complication after hematopoietic stem cell transplantation (HSCT). Gut is the most vulnerable target organ of acute GVHD. Patients who develope the acute gut GVHD and do not respond to the first line therapy with steroids have a high mortality. The investigation of safe and effective second line therapy for these patients are in need. The study evaluates safety and efficacy of fecal microbiota transplantation (FMT) for the treatment of streoid resistant GVHD of the gut. Stool for FMT will be prepared from the healthy donor.This strategy might offer a safe and effective therapeutic approach for these acute steroid resistant gut GVHD patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults(ages are elder than 18 years and younger than 75 years) who developed gut acute Graft-versus-Host Disease(aGVHD) after allogeneic hematopoietic stem cell transplantation(HSCT) and were resistant to a first line therapy with steroids.

  2. patients who were diagnosed as Stage 3 or 4 Gastro-intestinal Acute Graft-versus-Host(GI-aGVHD) with the symptoms such as diarrhea or abdominal pain.

  3. Participants who accepted the FMT treatment. 4. Signature of informed and written consent by the subject.

Exclusion Criteria:

* 1. patients who were diagnosed as Stage 1 or 2 Gastro-intestinal Acute Graft-versus-Host(GI-aGVHD) 2. patients with unstable vital signs or severe cardiac and pulmonary disorder. 3. patients who were failure to cooperate endoscopy examination. 4. patients who were younger than 18 years or pregnant. 5. patients who were poor compliance to FMT treatment. 6. patients who were not able to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Gut acute Graft-versus-Host Disease (aGvHD) response. | 1 day to 7 days following FMT
  Participants will be evaluated within 7 days following transplantation for response to therapy.

SECONDARY OUTCOMES:
Non-serious adverse events | 1,3,5,7 days following FMTs
  Participants will be evaluated for non-serious adverse events relating to FMT within 7 days following transplantation. Non-serious adverse events are defined as diarrhea, nausea and vomiting, fatigue and malaise, headache, and distension/bloating/abdominal discomfort/pain.
aGvHD severity | 1,3,5,7 days following FMT
  Number of participants will be evaluated on 1，3，5, 7 days following transplantation for severity of aGvHD.
Number of participants with infectious disorders | 1,3,5,7 days following FMT
  Evaluation of FMT activity on infectious disorder.
Number of multidrug resistant bacteria in faeces | 1,3,5,7 days following FMT
  Evaluation of FMT activity on multidrug-resistant bacteria (MDRB) carriage
Change in microbiota composition after FMT | 1,3,5,7 days months following FMT
  Evaluation of microbiota composition before and after FMT

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital to Academy of Military Medical Sciences, Beijing, Beijing Municipality, China